CLINICAL TRIAL: NCT05625737
Title: A Single-center, Single-arm, Open-label, Exploratory Study Evaluating Fruquintinib Combined with Sintilimab in Second-line Treatment of Patients with Advanced Gastric or Gastro-esophageal Junction Adenocarcinoma
Brief Title: Fruquintinib Combined with Sintilimab As Second-line Therapy for Gastric or Gastro-esophageal Junction Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hongli Liu, Director, Head of GI Department , Principal Investigator, Clinical Professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-CC-GC003
Record Dates: First submitted 2022-11-09; First posted 2022-11-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fruquintinib plus Sintilimab (Experimental): Fruquintinib combined with sintilimab. Fruquintinib: 4 mg/d, qd, po, d1-14, q3w; Sintilimab: 200 mg/d, ivgtt, d1, q3w.
  Interventions: Drug: Fruquintinib; Drug: Sintilimab

INTERVENTIONS:
Drug: Fruquintinib — Fruquintinib will be administrated as 4mg orally, once daily for 2 weeks on/1 week off.
Drug: Sintilimab — Sintilimab will be administrated as 200mg once every 3 weeks.

SUMMARY:
This was a single-arm, prospective study to investigate the efficacy and safety of fruquintinib combined with sintilimab in the second-line treatment of Chinese patients with advanced gastric/GEJ adenocarcinoma.

DETAILED DESCRIPTION:
Patients with adenocarcinoma of the gastro-esophageal junction or the stomach who have documented progression after being treated with a 1st line chemotherapy can be included. All patients will receive a second line therapy with fruquintinib and sintilimab, a checkpoint inhibitor. Clinical and radiographic assessment will be performed regularly. Patients will be treated until disease progression, untolerable toxicity or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Signed the Informed Consent Form
* Ages: 18-75 Years (concluding 18 and 75 Years)
* Pathologically confirmed unresectable advanced gastric/gastroesophageal junction adenocarcinoma
* Failure to 1st line therapy, completed at least 28 days before enrollment
* HER2-negative
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy greater than 3 months
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan, larger than 20 mm in diameter by conventional CT scan) according to RECIST1.1
* Sufficient organ functions as follows (any blood transfusion or cell growth factor use within 14 days before enrollment is not allowed):

Absolute Neutrophil Count (ANC) ≥1.5×109/L Platelet Count of ≥175×109/L; Hemoglobin≥90g/L; Total Bilirubin (TBIL) ≤1.5 x ULN; ALT and /or AST<1.5 x ULN; If there is liver metastasis, then ALT and/or AST<3.0 x ULN; Serum Creatinine (SCr) ≤1.5×ULN; Endogenous creatinine clearance rate ≥50ml / min；

* Man and woman who childbearing potential agrees to use adequate contraception
* Willingness to provide enough tumor tissues for PD-L1 expression test

Exclusion Criteria:

* Patients could not obey the study protocol.
* Previous therapy with VEGFR Inhibitor.
* Other malignancy within 5 years prior to study enrolment, except for cervical carcinoma in situ, basal or squamous cell skin cancer.
* Known brain or CNS metastases.
* Patients with any active autoimmune disease or a documented history of autoimmune disease within 4 weeks prior to enrollment.
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* Uncontrolled malignant ascites.
* Clinically significant cardiovascular diseases, including but not limited to acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Congestive heart failure, New York Heart Association (NYHA) grade > 2; ventricular arrhythmia requiring drug treatment; LVEF (left ventricular ejection fraction) < 50%.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Participation in another clinical trial with any experimental drug within 4 weeks prior to enrollment.
* Clinically significant electrolyte abnormalities judged by researchers.
* Systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg regardless of any antihypertensive drugs.
* Poorly controlled diabetes before enrollment.
* Any factors that influence the usage of oral administration and patients cannot take fruquintinib orally.
* Active gastric and duodenal ulcer, ulcerative colitis or uncontrolled hemorrhage in GI, or other conditions that may cause GI bleeding and perforation as determined by the investigator.
* Patients with obvious evidence of bleeding tendency or medical history within 3 months before enrollment, hemoptysis or thromboembolism within 12 months.
* Active infection or serious infection that is uncontrolled by drug (NCI CTCAE v. 5.0 Grade ≥ 2).
* History of clinically significant hepatic disease, including hepatitis B virus (HBV) infection with HBV DNA positive (copies ≥1×104/ml or >2000IU/ml); known hepatitis C virus infection with HCV RNA positive (copies ≥1×103/ml).
* Persisting toxicity related to prior therapy (NCI CTCAE v. 5.0 Grade > 1).
* Pregnant or breastfeeding female patient.
* Receive blood transfusion, blood products and hematopoietic factors such as albumin and granulocyte colony stimulating factor (G-CSF) within 14 days prior to enrollment.
* Other severe acute or chronic medical conditions including metabolic disorder, physical examination or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Urinary protein ≥ ++, and the 24-hour urine protein quantification is greater than 1.0 g.
* Use of immunosuppressive medication, or systemic/local immunosuppressive corticosteroids for complication.
* Patients considered unsuitable for inclusion in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | from date of randomization until the date of progressive disease or EOT due to any cause, assessed up to 1 year
  ORR is defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator.
Overall Survival (OS) | from date of randomization until the date of death due to any cause, assessed up to 2 years
  OS is defined as the time from randomization to death due to any cause.
Disease Control Rate (DCR) | from date of randomization until the date of progressive disease or EOT due to any cause, assessed up to 1 year
  DCR is defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
Duration of Response (DoR) | from date of the first documentation of response to the date of the first documentation of objective tumor progression or death due to any cause, whichever came first, assessed up to 1 year
  DoR is defined as the time how long response lasts
Adverse Event (AEs) | from the date of first dose to the 30 days post the last dose
  Safety will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.

OTHER OUTCOMES:
Exploratory endpoint | from date of randomization until the date of progressive disease or EOT due to any cause, assessed up to 1 year
  To identify the correlation between PD-L1 expression and inflammatory factor score with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Liu, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No